CLINICAL TRIAL: NCT04615377
Title: The Kaia hiP and Knee paIn Digital Application as an interVention for Self-management of Pain in Patients With OsteoarThritis - a Randomised Controlled Study (Kaia PIVOT Study).
Brief Title: The Kaia Hip and Knee Pain Intervention for Self-management of the Pain in Patients With Osteoarthritis.
Acronym: PIVOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaia Health Software (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kaia US OA Study; USOA001 (Other: Kaia Health Software, Inc.)
Record Dates: First submitted 2020-10-23; First posted 2020-11-04 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Knee Osteoarthritis; Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kaia hip and knee pain app (Experimental): Kaia software application: Kaia Knee and Hip pain app (version 2.37.0) The Kaia Knee and Hip pain app is an investigational device, which is intended as a digital aid for the self-management of osteoarthritis for use by adults (between 22 to 75 years old) without supervision by healthcare professionals in a home setting.
  Interventions: Behavioral: Kaia hip and knee pain application
- Treatment as usual (Active Comparator): Participants will be encouraged to continue the treatment that they have been on without restriction
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Kaia hip and knee pain application — The Kaia Knee and Hip pain app software, when loaded onto a smartphone, recommends to the participant specific exercises for the lower extremity. Using the camera on a smartphone, the software then tracks the participant's movements as the participant performs the exercises, analyzes those movements using machine learning, and provides audio-visual feedback to the participant. The exercise therapy is augmented by educational content and cognitive behavioral therapy to provide a multidisciplinary approach to self-management of osteoarthritis. Behavioral Health Coaches ensure participant motivation throughout the program based on a predefined curriculum.
  Arms: Kaia hip and knee pain app
Other: Treatment as usual — Participants allocated to the control arm will be advised to continue receiving treatment as usual ( standard care) without restrictions, except participation in other investigational trials, and will likewise be followed up for 90 days. Apart from that, they are encouraged to seek care, as they would do normally.
  Arms: Treatment as usual

SUMMARY:
The study intervention provides an innovative way of making exercise training and other recommended lifestyle modifications as accessible as possible for knee and hip OA participants by introducing a home-based exercise training program with a motion track feedback technology. Self-management of the pain for the patients suffering osteoarthritis, in the form of lifestyle modification, implementation of coping strategies and exercise is part of recommendations of recent international guidelines such as those by the Osteoarthritis Research Society International (OARSI). Cost and resource constraints typically limit the access to these recommended therapies. Moreover, the study intervention is focused on maintaining and adapting everyday physical activity, as required, in comparison to the control group.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a painful, degenerative disease of the affected joints. According to surveys by the World Health Organization (WHO) knee and hip joint OA is one of the diseases that make up the largest proportion of all disability diseases.

On the individual patient level, there is a pronounced limitation of the quality of life, which can also lead to the development of secondary diseases. There are numerous methods available for the treatment of OA, the spectrum of which ranges from conservative measures such as physical therapy or medical procedures up to surgical procedures, especially joint replacement. In recent years, the number of prostheses implanted in knee and hip joints has increased significantly.

International guidelines such as those of the American College of Rheumatologists recommend conservative treatment of OA of the knee and hip joint with physical therapy. Multidisciplinary approaches include aerobic and anaerobic exercise training, in particular with the aim of weight loss in overweight participants, participant education for self-management of the disease and the consideration of psychosocial factors. This comprehensive, structured, conservative program for the treatment of OA achieves significantly better results than the standard treatment. However, comparable programs, which offer comprehensive management of OA are not widely available.

Digital therapies represent a novel approach to help patients manage themselves and their diseases in a home setting and even show better results than current standard therapies. An analysis of a smartphone intervention providing a multidisciplinary approach for self-management of lower back pain, the Kaia Back Pain Relief app, shows promising results in 180 users with a significant and clinically relevant reduction of pain levels.

Based on these promising results, this study will evaluate the effectiveness of the Kaia Knee and Hip pain app intervention in comparison to usual medical care in reducing pain and disease-related symptoms in participants with OA over 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Between 22 and 75 years old
* Able to speak, read, and understand English
* Able to use an iPad, has internet access at home and a personal email address
* Self-reported diagnosis of OA of knee or hip confirmed by ACR clinical criteria
* Self-reported pain intensity ≥4/10 on Numeric Rating Scale (NRS) for knee and hip pain, on average, in the week prior to screening
* Pain duration ≥1 month
* Willing and capable of providing Informed Consent to use the Kaia Knee and Hip pain app and participate in all assessments associated with this clinical study

Exclusion Criteria:

* Referral or plans for surgery, chiropractic care, acupuncture, physical therapy, injections or other treatment for knee or hip pain in the next 3 months following screening
* Self-reported prior subscription to Kaia apps or plans to participate in any other investigational trials or protocols for knee or hip pain
* Prior knee or hip surgery or injury in the last 3 months
* Current workers comp case or litigation related to musculoskeletal pain
* Self-reported use of opioids within 30 days prior to screening
* Self-reported history of substance abuse within the past 1 year
* Self-reported diagnosis of an inflammatory/rheumatologic disease
* Self-reported diagnosis of neuropathic pain disorder or other chronic pain disorder (ex. fibromyalgia, complex regional pain syndrome [CRPS])

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index as calculated from Hip disability and Osteoarthritis Outcome Score (HOOS) or Knee injury and Osteoarthritis Outcome Score (KOOS). | On day 0, 30, 60 and 90
  The primary endpoint is to evaluate the change in the Western Ontario and McMaster Universities Osteoarthritis Index as calculated from Hip disability and Osteoarthritis Outcome Score (HOOS) or Knee injury and Osteoarthritis Outcome Score (KOOS).This change will be calculated over day 0 until week 12. Where the higher scores on the HOOS and KOOS indicate worse pain, stiffness, and functional limitations. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).

SECONDARY OUTCOMES:
Pain index as in western Ontario and McMaster's Osteoarthritis Index as derived from Hip disability and Osteoarthritis Outcome Score (HOOS) or Knee injury and Osteoarthritis Outcome Score (KOOS). | On day 0, 30, 60 and 90
  To evaluate the change from baseline by Hip disability and Osteoarthritis Outcome Score (HOOS) or Knee injury and Osteoarthritis Outcome Score (KOOS) and derive the pain score for the Western Ontario and McMaster Universities Osteoarthritis Index pain sub-scale through Week 12 i.e pain score domain (mean of changes in the 5 pain related items) on HOOS or KOOS. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
Functionality index as in western Ontario and McMaster's Osteoarthritis Index as derived from Hip disability and Osteoarthritis Outcome Score (HOOS) or Knee injury and Osteoarthritis Outcome Score (KOOS). | On day 0, 30, 60 and 90
  To evaluate the change from baseline by Hip disability and Osteoarthritis Outcome Score (HOOS) or Knee injury and Osteoarthritis Outcome Score (KOOS) and derive the Functionality index as for the Western Ontario and McMaster Universities Osteoarthritis functionality sub-scale through Week 12 i.e pain score domain (mean of changes in the 5 pain related items) on HOOS or KOOS. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
Stiffness score as in western Ontario and McMaster's Osteoarthritis Index as derived from Hip disability and Osteoarthritis Outcome Score (HOOS) or Knee injury and Osteoarthritis Outcome Score (KOOS). | On day 0, 30, 60 and 90
  To evaluate the change of stiffness from baseline, by Hip disability and Osteoarthritis Outcome Score (HOOS) or Knee injury and Osteoarthritis Outcome Score (KOOS), and derive the stiffness index score as for the Western Ontario and McMaster Universities Osteoarthritis stiffness sub-scale, through Week 12 i.e stiffness score domain (mean of changes in the 5 pain related items) on HOOS or KOOS. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
Patient-Reported Outcomes Measurement Information System (PROMIS Global 10) | Information collected on day 0, 30, 60 and 90
  Overall change in the Quality of life score assessed by the PROMIS Global 10 questionnaire from baseline to the week 12.
Inclination towards healthcare utilization | Information collected only on day 0
  Self-reported inclination towards healthcare utilization on an 11-point Likert scale. Where (0) means none and (11) means Extreme.
Self-reported number of lost workdays | Information collected only on day 0 and day 90
  Self-reported number of lost workdays in the month prior to enrolment and during study observational period (assessed at baseline day 0, day 30, day 60, and day 90)
Pain medication intake | Information collected on day 0, 30, 60 and 90
  Pain medication intake 30 days prior to enrolment and during study period.

OTHER OUTCOMES:
Perceived treatment helpfulness | Study start, On day 0
  Feedback on the mobile medical application (5-Point Likert Scales ranging from 1 "lowest satisfaction" to 5 "highest satisfaction")
Satisfaction and perceived treatment helpfulness | Study end, On day 90
  Feedback on the mobile medical application (5-Point Likert Scales ranging from 1 "lowest satisfaction" to 5 "highest satisfaction")
Self-reported healthcare utilization | On day 0, 30, 60 and 90
  Use of services by persons for the purpose of preventing and curing health problems (type and number of times utilized)
Safety assessment | On day 0, 30, 60 and 90
  The safety of the usage of the Kaia Knee and Hip pain app is evaluated by the incidence of reported adverse events in the intervention and control arm.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Choo, MD, Principal Investigator — Orthopaedic and Neurosurgery Specialists, 6 Greenwich Office Park, Greenwich, CT 06831
Locations (1):
- Choo, Stamford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No